CLINICAL TRIAL: NCT00793117
Title: The Evaluation of Effect of Pva Sponge in Prevention of Complications in Fess
Brief Title: The Effect of Packing in Post Operative Management of FESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Babak Saedi, associate Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BS-87-01-48-6841; 87-01-48-6844
Record Dates: First submitted 2008-11-15; First posted 2008-11-19 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Epistaxis; Nasal Obstruction; Pain
Keywords: chronic sinusitis; FESS; packing
MeSH Terms: conditions — Epistaxis; Nasal Obstruction; Pain | interventions — Drug Packaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): poly vinil chloride packing
  Interventions: Procedure: packing

INTERVENTIONS:
Procedure: packing — packing in middle meatus for duration of 5 day

SUMMARY:
Chronic sinusitis is a very common problem. The functional endoscopic sinus surgery is a prevalent option to treat this disease.During usage of different techniques of surgery, the need for packing after surgery is debatable problem. So to solve this problem this research has been designed.

DETAILED DESCRIPTION:
Chronic sinusitis is a very common problem. The functional endoscopic sinus surgery is a prevalent option to treat this disease.During usage of different techniques of surgery, the need for packing after surgery is debatable problem.

Someone claimed packing is unnecessary and other one propose different material to packing after surgery. So to solve this problem this research has been designed.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic sinusitis who candid of fess

Exclusion Criteria:

* Systemic disease
* Corticosteroid usage counterindication
* Immune suppresive usage
* Choncha bollusa resection-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
complication | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: babak saedi, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Imam Khomaimee hospital, Tehran, Tehran Province, Iran